CLINICAL TRIAL: NCT03475563
Title: BiOSS LIM C Stent Registry in Bifurcated Lesions
Brief Title: BiOSS Study (BiOSS LIM C Stent Registry in Bifurcated Lesions)
Acronym: BIOSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BIOSS
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stent; Dedicated bifurcation stent; Cobalt-chromium; Sirolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with coronary artery disease: (coronary artery disease)
  Interventions: Procedure: Coronary angioplasty with stent implantation

INTERVENTIONS:
Procedure: Coronary angioplasty with stent implantation — Coronary angioplasty with BiOSS LIM C stent implantation

SUMMARY:
The BIOSS Lim C pharmacoactive Stent has characteristics of design that makes it very suitable for the treatment of bifurcational lesions . The objective of the study is providing deeper knowledge into the results of this stent in the treatment of bifurcational lesions.

DETAILED DESCRIPTION:
The BIOSS Lim C pharmacoactive Stent has characteristics of design that makes it very suitable for the treatment of bifurcational lesions . The objective of the study is providing deeper knowledge into the results of this stent in the treatment of bifurcational lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Clinical indication of coronary angioplasty in bifurcated lesion.
* Bifurcated lesions with both distal branches at least 2 mm in diameter.
* The lesion must be located in the main branch, with a severe stenosis by visual estimation at some point in the main branch, with or without involvement of the lateral branch.
* Express acceptance and signature of informed consent.

Exclusion Criteria:

* Express rejection of the patient to participate in the study.
* Exclusive involvement of the lateral branch (Medina lesion 001).
* Contraindication for antiplatelet treatment.
* Lesions due to restenosis.
* Lesions in saphenous grafts.
* Total chronic occlusions.
* Cardiogenic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease referred for coronary revascularization will be included with susceptible lesion of coronary intervention in bifurcation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Successful angioplasty | 1 day
  After angiography: TIMI (thrombolysis in myocardial infarction ) 3 (both branches). With respect to reference diameter, none of the segments treated with stent has a residual stenosis> 30% or> 50% in those not treated with stent.
MACE | 30 days
  Cumulative rate of major adverse cardiovascular events (MACE) including cardiac death, myocardial infarction (MI) and repeated revascularization of the target lesion (TLR)
MACE | 1 year
  Cumulative rate of major adverse cardiovascular events (MACE) including cardiac

SECONDARY OUTCOMES:
Target vessel revascularization | 30 days
  Target vessel revascularization
Percentage of stent struts malposition | 30 days
  Percentage of stent struts malposition
contrast media volume | 1 day
  contrast media volume
Angioplasty time | 1 day
  Angioplasty time

CONTACTS AND LOCATIONS:
Overall Officials: Imanol Otaegui, MD, Principal Investigator — Hospital Universitari Vall d'hebron Barcelona, Spain
Locations (3):
- Spain (3):
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de León, León

REFERENCES:
- [Result] Gil RJ, Bil J, Dzavik V, Vassilev D, Kern A, Formuszewicz R, Zalewska-Adamiec M, Dobrzycki S. Regular Drug-Eluting Stent vs Dedicated Coronary Bifurcation BiOSS Expert Stent: Multicenter Open-Label Randomized Controlled POLBOS I Trial. Can J Cardiol. 2015 May;31(5):671-8. doi: 10.1016/j.cjca.2014.12.024. Epub 2014 Dec 24. PMID 25828372
- [Result] Gil RJ, Bil J, Vassiliev D, Inigo Garcia LA. First-in-man study of dedicated bifurcation sirolimus-eluting stent: 12-month results of BiOSS LIM(R) Registry. J Interv Cardiol. 2015 Feb;28(1):51-60. doi: 10.1111/joic.12180. PMID 25689548
- [Result] Gil RJ, Bil J, Grundeken MJ, Inigo Garcia LA, Vassilev D, Kern A, Pawlowski T, Wykrzykowska JJ, Serruys PW. Long-term effectiveness and safety of the sirolimus-eluting BiOSS LIM(R) dedicated bifurcation stent in the treatment of distal left main stenosis: an international registry. EuroIntervention. 2016 Nov 20;12(10):1246-1254. doi: 10.4244/EIJY15M10_05. PMID 26465375